CLINICAL TRIAL: NCT04739605
Title: Postoperative Patient-reported Quality of Recovery in Colorectal Surgery Patients Under Enhanced Recovery After Surgery Program Using QoR-15.
Brief Title: Quality of Recovery Using QoR-15 in Enhanced Recovery After Colorectal Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of the Anesthesiology department, University of Liege
Other Study IDs: 2021-colorectal-QoR15
Record Dates: First submitted 2021-02-03; First posted 2021-02-04 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Surgery; Patient-related Outcomes Measures; Enhanced Recovery After Surgery
Keywords: colorectal; enhanced recovery; patient-related outcomes measures; QoR15

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will evaluate the patient reported outcomes and postoperative patient-related quality of recovery in 150 patients undergoing colorectal surgery within an enhanced recovery program at CHU Liège. The QoR15 survey will be performed preoperatively and repeated postoperatively at hospital or via telephone calls on Day + 1, Day +2; Day + 3, Day 7 and Day + 14. The total score and the score at the subsections will be correlated with the medical and surgical characteristics of the patients.

DETAILED DESCRIPTION:
For several years, we have been applying the concept of Enhanced Recovery Program (ERP) for colorectal surgery at CHU Liége (Belgium). Since October 2015, the University Hospital of Liège has been labelled as reference center for ERP after colorectal surgery by a French-speaking organization GRACE (French-speaking group for Enhanced Recovery after Surgery; www.grace-asso.fr). Despite the benefits for the patient and the economic benefits of such programs, few studies have investigated postoperative patient-related quality of recovery of patients who have had ERP.

This observational study will evaluate the patient reported outcomes and postoperative patient-related quality of recovery in 150 patients undergoing colorectal surgery according to an ERP at CHU Liège.The QoR15 survey will be performed preoperatively and repeated postoperatively at hospital or via telephone calls on Day + 1, Day +2; Day + 3, Day 7 and Day + 14. The total score and the answers at the subsections will be correlated with the medical and surgical characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* •any patient scheduled for colorectal surgery within an ERP at CHU Liège
* Correct comprehension of french

Exclusion Criteria:

* •unable to answer the survey (cognitive disorders, bad knowledge of the French language)
* •closure of loop ileostomy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient schedules for colorectal surgery with the ERP at CHU Liège (Belgium). Patients age must be greater than 18 years. There is no maximum limit of age.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Difference of Quality of recovery-15 (QoR-15) score between the preoperative scopre at Day 0 and postoperative score at Day 1 and its link between length of stay and occurrence of complication. | 2 weeks
  The score of the Quality of recovery-15 (QoR-15) Survey and subscores. The 11-point numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Brichant, PhD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU de Liege, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No